CLINICAL TRIAL: NCT00011544
Title: Physical Performance Measures for Manual Wheelchair Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: B1751R
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Spinal Cord Injury
Keywords: wheelchair, biomechanics, aging, functional outcome, disability
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: Performance Measure

SUMMARY:
The project is intended to modify the Functional Independence Measure (FIM) for manual wheelchair users. It will determine if the new measure is a better measure of community independence for manual wheelchair users than the FIM. During the Phase 1 of the study it will then use this new measure to determine whether a home exercise program increases functional independence in wheelchair users. In Phases II and III of the study 120 manual wheelchair users will participate to test and validate the new measure and to test the effectiveness of therapeutic exercise. Subjects will range in age from 20 to 79 yrs. and have a variety of disabilities.

ELIGIBILITY:
Wheelchair users

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1998-01; Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D., Asst. Director — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Baltimore, Baltimore, Maryland, United States